CLINICAL TRIAL: NCT06152627
Title: Towards a Unified System to Classify Treatments for Muscle Tension Dysphonia
Brief Title: Voice Therapy Per the Rehabilitation Treatment Specification System
Acronym: RTSS-Voice
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Emory University (Other); New York University (Other); University of Utah (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Jarrad Van Stan, Associate Professor of Surgery and Speech-Language Pathology, Massachusetts General Hospital
Other Study IDs: 2023P003127
Record Dates: First submitted 2023-11-19; First posted 2023-11-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Muscle Tension Dysphonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- First Year of RTSS-Voice use: These 300 patients from five Voice Centers will receive standard of care voice therapy where their treating clinicians will be trained to use the RTSS-Voice in their documentation.
  Interventions: Behavioral: Standard of care voice therapy with novice clinician RTSS-Voice documentation
- Second Year of RTSS-Voice use: These 300 patients from five Voice Centers will receive standard of care voice therapy where their treating clinicians have already been trained to use the RTSS-Voice in their documentation.
  Interventions: Behavioral: Standard of care voice therapy with expert clinician RTSS-Voice documentation

INTERVENTIONS:
Behavioral: Standard of care voice therapy with novice clinician RTSS-Voice documentation — Voice therapy is individually tailored to each patient and typically includes behavioral ingredients (e.g., applying pressure to the anterior neck, practice voicing in various ways, feedback on performance, provide information on the importance of therapy concepts) to modify the patient's auditory, somatosensory, vocal, musculoskeletal, respiratory, and mental functions. During this time, the treating clinicians will be trained to use the RTSS-Voice in their clinical documentation.
  Groups: First Year of RTSS-Voice use
Behavioral: Standard of care voice therapy with expert clinician RTSS-Voice documentation — Voice therapy is individually tailored to each patient and typically includes behavioral ingredients (e.g., applying pressure to the anterior neck, practice voicing in various ways, feedback on performance, provide information on the importance of therapy concepts) to modify the patient's auditory, somatosensory, vocal, musculoskeletal, respiratory, and mental functions. During this time, the treating clinicians will have completed their RTSS-Voice training and using the RTSS-Voice in their clinical documentation.
  Groups: Second Year of RTSS-Voice use

SUMMARY:
The goal of this study is to evaluate if using evidence-based, standard ingredient and target codes from the Rehabilitation Treatment Specification System - Voice Therapy (RTSS-Voice) in standard of care voice therapy documentation can improve outcomes for patients with muscle tension dysphonia (MTD). The main question it aims to answer is: Since the RTSS-Voice will help clinicians think about their treatment more specifically and in relation to nine evidence-based therapies, will its adoption be associated with improved outcomes? Clinicians across five voice centers will be asked to use the RTSS-Voice to document their voice therapy sessions for patients with MTD. Researchers will compare changes in outcomes between two groups of patients: those treated during the clinician's first year using the RTSS-Voice versus those treated during the clinician's second year using the RTSS-Voice.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if using evidence-based, standard ingredient and target codes from the Rehabilitation Treatment Specification System - Voice Therapy (RTSS-Voice) in standard of care voice therapy documentation can improve outcomes for patients with muscle tension dysphonia (MTD). RTSS-Voice adoption is likely to be associated with improved outcomes because it requires clinicians to think about their therapy in relation to nine evidence-based therapies (i.e., increased evidence-based practice) and more carefully consider the specific changes in targets directly related to specific clinical actions, i.e., improved clinical reasoning. Sixty patents will be enrolled per year (at minimum) from each of the five participating voice centers, i.e., 300 patients in Years 1 and 2 (total patients = 600). For each patient, outcomes will be collected before and after therapy including patient-reported vocal functioning, clinician-reported voice quality, an objective measure associated with overall voice quality (Cepstral Peak Prominence/CPP), and total number of sessions. Each voice center uses different patient-reported and clinician-reported measures. Thus, linear regression models will examine changes in outcomes during Year 1 versus Year 2 for each individual site. The different patient- and clinician-reported measures have been found to be highly correlated. Therefore, individual sites will also be pooled together in a mini meta-analysis. Standardized effect sizes (Cohen's d) will be calculated for each site, representing the effect of RTSS-Voice adoption. Using a fixed effects model, an average effect size across sites will be calculated, weighted by sample size. The average effect size across sites will then represent the overall effect of the implementation on vocal functioning, voice quality, CPP, and number of sessions. Power: The investigators anticipate a minimum of 60 patients per site, (total of 300 patients per year). For site-specific analyses, a sample size of 60 patients for each group (Year 1 versus Year 2) is associated with 80% power to detect the smallest clinically meaningful effect size: d = .5. The effect size d = .5 was chosen because it is the smallest effect that is "visible to the naked eye" associated with rejecting the null hypothesis and supporting the alternative hypothesis in rehabilitation treatment studies and used in multiple voice studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Muscle Tension Dysphonia (pMTD)
* Patients with pMTD will be included regardless of subtype (e.g., functional aphonia, vocal fry, ventricular dysphonia) and they can have secondary diagnoses of reflux.

Exclusion Criteria:

* Patients diagnosed with pMTD will be excluded if they have secondary diagnoses related to structural, neurological, or respiratory disorders such as laryngitis, obvious vocal fold nodules, polyps, cyst, granuloma, sulci, paradoxical vocal fold motion, chronic cough, confirmed or possible upper airway paralysis/paresis, dysphagia, polypoid corditis, keratosis, presbylarynx, leukoplakia, or history of radiation to the head/neck. Patients with pMTD will be included regardless of subtype (e.g., functional aphonia, vocal fry, ventricular dysphonia) and they can have secondary diagnoses of reflux.
* Non-English speakers. The RTSS-Voice's standard and operationalized categories are in English.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All recruited patients will be diagnosed with primary Muscle Tension Dysphonia (pMTD) because: [1] clinical impact - pMTD is the most commonly treated voice disorder; [2] minimal diagnostic confounds - pMTD is ostensibly behavioral (i.e., no variations in disordered anatomy/physiology) and voice therapy is the only curative option (i.e., minimal presence of other treatments like sur-gery); [3] comprehensive coverage of therapy concepts - pMTD is the most heterogeneous voice disorder; [4] availability of multiple therapies with similar outcomes - allowing us to use previously developed methods for identifying unique targets/ingredients.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Voice Health Index (VHI) | pre-intervention and immediately after the intervention
  The VHI consists of 30 Likert questions ranging from 0-4 (0 = never, 1 = almost never, 2 = sometimes, 3 = almost always, 4 = always) that estimate how the patient's vocal function effects his/her daily life. A short-form can be used (the VHI-10) that uses a subset of 10 questions from the 30 total questions. This patient-reported outcome measure will be used to evaluate if the patients perceive that therapy helped them function better in their activities of daily living.
Voice-Related Quality of Life (V-RQOL) | pre-intervention and immediately after the intervention
  The V-RQOL consists of 10 Likert-style questions ranging from 1-5 (1 = none not a problem at all, 2 = a small amount, 3 = a moderate (medium) problem, 4 = a lot, 5 = problem is "as bad as it can be") that estimate how the subject's vocal function effects his/her daily life. This patient-reported outcome measure will be used to evaluate if the patients perceive that therapy helped them function better in their activities of daily living.
Consensus Auditory Perceptual Evaluation of Voice (CAPE-V) | pre-intervention and immediately after the intervention
  The CAPE-V consists of 4 perceptually judged 100-mm visual analog scales (Overall dysphonia, Breathiness, Strain, Roughness). The patient's treating voice specialized speech-language pathologist will judge the audio samples. These judgements provide gold-standard, perceptual ratings of voice quality to evaluate if voice therapy is associated with improved voice quality.
Grade Roughness Breathiness Asthenia Strain (GRBAS) Scale | pre-intervention and immediately after the intervention
  The GRBAS consists of 5 perceptually-judged scales (Grade, Roughness, Breathiness, Asthenia, Strain) on a 0-3 Likert scale (0 = normal, 1 = mild severity, 2 = moderate severity, 3 = severe). The patient's treating voice specialized speech language pathologist will judge the audio samples. These judgements provide gold-standard, perceptual ratings of voice quality to evaluate if voice therapy is associated with improved voice quality.
Cepstral Peak Prominence (CPP) | pre-intervention and immediately after the intervention
  To calculate CPP, all voiced 50 millisecond (ms) frames will undergo two discrete Fourier transforms computed in succession with a logarithmic transformation between them. A regression line is then computed over quefrencies greater than 2 ms (corresponding to a quefrency range minimally affected by subglottal resonances). Finally, the CPP for each frame is defined as the difference, in decibels (dB), between the magnitude of the highest peak and the baseline regression level in the power cepstrum. The peak search is limited to quefrencies between 2.5 ms and 12 ms, corresponding to frequencies of 417 Hertz (Hz) and 83 Hz, respectively. The resulting CPP is an estimate of periodicity in the voice signal, which has strongly correlated to overall dysphonia in multiple previous studies. This will be used to quantitatively evaluate if voice therapy was associated with improved overall voice quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jarrad Van Stan, PhD, CCC-SLP, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University, New York, New York
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
We expect to share de-identified data on the 600 patients before and after therapy. Specifically, changes in patient-reported outcomes, clinician-reported outcomes, an objective measure of periodicity, and number of therapy sessions.
Supporting Information: Study Protocol, SAP
Time Frame: Data collection will be finished by August 2027. Since the data is de-identified at time of data collection, we will plan to submit the data as soon as possible to a generalist repository approved by the PI's home institution and meets all National Institutes of Health Generalist Repository requirements: Harvard Dataverse. The National Institute on Deafness and Other Communication Disorders participates in multiple domain specific repositories (aphasia, fluency, multiple brain repositories, mice work, and Downs syndrome). However, there are no domain-specific repositories for voice, voice disorders, or motor control/learning data.
Access Criteria: The study datasets will be collected with the following informed consent: Health/Medical/Biomedical. To maximize the appropriate sharing of scientific data and protect research participants' privacy and confidentiality, reuse of this dataset should use the following Data Use Limitations under Controlled Access that is made available by a data repository only after approval of the request by the Harvard Dataverse independent review panel process.